CLINICAL TRIAL: NCT05302128
Title: The Effect of Cold Vapor on Nausea and Vomiting in the Early Postoperative Period After Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Atlas University (Other)
Responsible Party: Principal Investigator, Dr. Özlem İbrahimoğlu, Assisstant Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IstanbulMU12
Record Dates: First submitted 2022-03-07; First posted 2022-03-31 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Laparoscopic Cholecystectomy; Postoperative Nausea; Postoperative Vomiting
Keywords: Nausea; Vomiting; Nursing care
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: Patients who were hospitalized for laparoscopic cholecystectomy and met the sample selection criteria will be included in the experimental and control groups by block randomization method using the random numbers table on the computer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold vapor group (Experimental): Cold vapor will be applied to the experimental group patients for 15 minutes in the recovery room. For the study, Nebtime UN600A Ultrasonic Nebulizer Device will be used to apply cold steam to the patients which used in the hospital and calibrated (https://elmaslarmedikal.com.tr/urunler/nebtime-un600aultrasonik-nebulizator/). The parameters to be set on the device for the cold vapor to be applied to the patients in the early postoperative period will be vapor intensity level 5 (1-10), air blowing intensity 5 (1-10), heater intensity 1 (+10C), and timer 15 minutes. The patients will be evaluated by the researchers in terms of nausea and vomiting before and 15 minutes after the cold vapor application in the recovery room and at the 2nd, 6th, 12th, and 24th hours after the cold vapor application in the postoperative service.
  Interventions: Other: Cold vapor
- Control group (No Intervention): Patients in the control group will receive standard care that includes all medical and non-medical treatments in the hospital. Nursing care, which is routinely applied to patients in the postoperative period, both in the recovery room and in the service, will be continued within the standard care. The patients will be evaluated by the researchers in terms of nausea and vomiting when they come to the recovery room and at the 2nd, 6th,12th, and 24th hours after the surgery in the postoperative service.

INTERVENTIONS:
Other: Cold vapor — Before surgery, the socio-demographic data of the patients will be recorded. After surgery, patients will be evaluated in the recovery room for their suitability to participate in the study with the Ramsay sedation scale and the Modified Aldrete Scale. Cold vapor will be applied to the patients for 15 minutes in the recovery room during the postoperative period. The parameters to be set on the device for the cold vapor to be applied to the patients in the early postoperative period will be vapor intensity level 5, air blowing intensity 5, heater intensity 1 (+10C), and timer 15 minutes. The patients will be evaluated by the researchers in terms of nausea and vomiting before and 15 minutes after the cold vapor application in the recovery room and at the 2nd, 6th,12th, and 24th hours after the cold vapor application in the postoperative service.
  Arms: Cold vapor group

SUMMARY:
Postoperative nausea and vomiting (PONV) was defined by the American Society of PeriAnesthesia Nurses (ASPAN) as nausea and/or vomiting in the first 24 hours after surgery and is among the most common complications after pain in patients undergoing surgery. PONV is divided into three as early, late, and delayed. Nausea-vomiting developing within 2-6 hours after surgery is classified as early, nausea-vomiting developing within 6-24 hours after surgery is classified as delayed, and nausea and/or vomiting developing within the first 24 hours after surgery are classified as delayed PONV. PONV increases the length of stay in the recovery room, delays starting oral intake, causes fluid and electrolyte imbalance, and causes pain, dehydration, delayed wound healing, decreased patient comfort, prolonged hospitalization, and increased cost. Therefore, the prevention and management of nausea and vomiting in the perioperative period in surgical patients are very important.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) was defined by the American Society of PeriAnesthesia Nurses (ASPAN) as nausea and/or vomiting in the first 24 hours after surgery and is among the most common complications after pain in patients undergoing surgery. PONV increases the length of stay in the recovery room, delays starting oral intake, causes fluid and electrolyte imbalance, and causes pain, dehydration, delayed wound healing, decreased patient comfort, prolonged hospitalization, and increased cost. Therefore, the prevention and management of nausea and vomiting in the perioperative period in surgical patients are very important.

In a meta-analysis study that included data from eleven countries, the prevalence of PONV was 27.7%, the prevalence of postoperative nausea was 31.4% and the prevalence of post-operative vomiting was 16.8%. In a study conducted in Turkey, it was reported that 45.9% of surgical patients had nausea and 23.6% had vomiting in the postoperative period. In another study conducted in the postoperative recovery unit, it was reported that 29% of the patients experienced nausea and vomiting.

The risk of PONV may vary depending on the patient, anesthesia, and surgical intervention. Patient-related risk factors include female gender, young age (under 50 years of age), obesity, history of motion sickness; anesthesia-related risk factors include the type of anesthesia, duration of administration, use of volatile anesthetics, opioids, and nitrous oxide; Among the risk factors for previous surgical interventions are laparoscopic, bariatric, gynecological and cholecystectomy surgeries.

Pharmacological treatment, non-pharmacological treatment methods, or both are used in the management of PONV in patients undergoing surgical intervention. Today, a multimodal approach is recommended in the management of PONV in early recovery protocols in surgical patients. Antiemetic drugs used among pharmacological methods can cause side effects such as headache, constipation, drowsiness, tremor, irregular heartbeat, and wound infection. Therefore, non-pharmacological treatment methods have an important place in care practices. In the literature, there are many studies on the successful application of non-pharmacological treatment methods such as massage, progressive relaxation exercises, hypnosis, acupuncture, yoga, acupressure, transcutaneous electrical nerve stimulation, music therapy, herbal treatments, and aromatherapy in the prevention of PONV.

The cold application creates vasoconstriction in the vessels in the area where it is applied, decreases the metabolic rate, and reduces edema. The cold application reduces muscle temperature by reducing the tension sensitivity of muscle spindles with the reflex effect of heat receptors or inactivating trigger points in the muscles and helps to reduce muscle spasm. Thus, it reduces skin sensitivity by lowering the temperature of nerve fibers and receptors. Cold application is especially beneficial in post-traumatic pain, swelling, and muscle spasm. Temperature can affect the release of odorous volatile substances in drugs. The cold application also has clinically important potential effects on nausea caused by unpleasant tastes by reducing the olfactory component of negative aromas. Cold can be applied in different ways. One of them is administration by inhalation. In the literature, there are studies on the positive effects of cold vapor application on sore throat, cough, swallowing, and hoarseness. In a study, it was determined that postoperative nausea and vomiting were less in patients who received oral care with the cold application after laparoscopic myomectomy compared to the control group. There is no study in the literature examining the effect of cold vapor application on PONV.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* To undergo laparoscopic cholecystectomy
* Having an ASA score of 1-2
* Getting 2 points from the Ramsay Sedation Scale in the postoperative recovery room.
* Having a Modified Aldrete score of at least 9 in the postoperative recovery room
* To be willing to participate in the study.

Exclusion Criteria:

* To undergo emergency surgery
* Being under the age of 18
* Having an ASA score of 3 and above
* Not agreeing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-04-11 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Cold vapor | First 24 hours after surgery
  The Visual Analogue Scale (VAS) of the patients for nausea who underwent cold vapor is decreased compared to those who do not. A score between 0 and 10 is taken from the VAS. It is good that the score from the VAS has decreased.
Cold vapor | First 24 hours after surgery
  The Postoperative Nausea and Vomiting Impact Scale of the patients for nausea and vomiting who underwent cold vapor are decreased compared to those who do not. A score between 0 and 6 is taken from the Postoperative Nausea and Vomiting Impact Scale. It is good that the score from the Postoperative Nausea and Vomiting Impact Scale has decreased.

IPD SHARING:
Plan to Share IPD: Undecided
A decision will be made after consultation with other researchers.

REFERENCES:
- [Background] Amirhosseini M, Dehghan M, Mangolian Shahrbabaki P, Pakmanesh H. Effectiveness of Aromatherapy for Relief of Pain, Nausea, and Vomiting after Percutaneous Nephrolithotomy: A Randomized Controlled Trial. Complement Med Res. 2020;27(6):440-448. doi: 10.1159/000508333. Epub 2020 Jun 23. PMID 32575103
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] American Society of PeriAnesthesia Nurses PONV/PDNV Strategic Work Team. ASPAN'S evidence-based clinical practice guideline for the prevention and/or management of PONV/PDNV. J Perianesth Nurs. 2006 Aug;21(4):230-50. doi: 10.1016/j.jopan.2006.06.003. No abstract available. PMID 16935735
- [Background] Boogaerts JG, Vanacker E, Seidel L, Albert A, Bardiau FM. Assessment of postoperative nausea using a visual analogue scale. Acta Anaesthesiol Scand. 2000 Apr;44(4):470-4. doi: 10.1034/j.1399-6576.2000.440420.x. PMID 10757584
- [Background] Brems C, Barnett J, Parret VC, Metzger J, Johnson ME. Alternative and complementary treatment needs and experiences of women with breast cancer. J Altern Complement Med. 2013 Jul;19(7):657-63. doi: 10.1089/acm.2012.0161. Epub 2013 Feb 1. PMID 23373443
- [Background] Bulut H, Erden S, Demir SG, Cakar B, Erdogan Z, Demir N, Ay A, Aydin E. The Effect of Cold Vapor Applied for Sore Throat in the Early Postoperative Period. J Perianesth Nurs. 2016 Aug;31(4):291-7. doi: 10.1016/j.jopan.2014.10.005. Epub 2016 Feb 24. PMID 27444760
- [Background] Campos de Carvalho E, Martins FT, dos Santos CB. A pilot study of a relaxation technique for management of nausea and vomiting in patients receiving cancer chemotherapy. Cancer Nurs. 2007 Mar-Apr;30(2):163-7. doi: 10.1097/01.NCC.0000265007.87311.d0. PMID 17413783
- [Background] Cronin SN, Odom-Forren J, Roberts H, Thomas M, Williams S, Wright MI. Effects of Controlled Breathing, With or Without Aromatherapy, in the Treatment of Postoperative Nausea. J Perianesth Nurs. 2015 Oct;30(5):389-97. doi: 10.1016/j.jopan.2015.03.010. PMID 26408513
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Background] Gecit S, Ozbayir T. Evaluation of Preoperative Risk Assessment and Postoperative Nausea and Vomiting: Importance for Nurses. J Perianesth Nurs. 2020 Dec;35(6):625-629. doi: 10.1016/j.jopan.2020.04.006. Epub 2020 Aug 7. PMID 32778493
- [Background] Gonella S, Dimonte V. Potential effects of pleasant and cold stimuli on nausea and vomiting induced by disgusting tastes. J Neurosci Res. 2016 May;94(5):366-77. doi: 10.1002/jnr.23724. Epub 2016 Feb 19. PMID 26896189
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Horn CC, Wallisch WJ, Homanics GE, Williams JP. Pathophysiological and neurochemical mechanisms of postoperative nausea and vomiting. Eur J Pharmacol. 2014 Jan 5;722:55-66. doi: 10.1016/j.ejphar.2013.10.037. Epub 2013 Oct 26. PMID 24495419
- [Background] Hunt K, Ernst E. The evidence-base for complementary medicine in children: a critical overview of systematic reviews. Arch Dis Child. 2011 Aug;96(8):769-76. doi: 10.1136/adc.2009.179036. Epub 2010 Jul 6. PMID 20605859
- [Background] Karagozoglu S, Tekyasar F, Yilmaz FA. Effects of music therapy and guided visual imagery on chemotherapy-induced anxiety and nausea-vomiting. J Clin Nurs. 2013 Jan;22(1-2):39-50. doi: 10.1111/jocn.12030. Epub 2012 Nov 8. PMID 23134272
- [Background] Karaman S, Karaman T, Tapar H, Dogru S, Suren M. A randomized placebo-controlled study of aromatherapy for the treatment of postoperative nausea and vomiting. Complement Ther Med. 2019 Feb;42:417-421. doi: 10.1016/j.ctim.2018.12.019. Epub 2018 Dec 28. PMID 30670276
- [Background] Kori K, Oikawa T, Odaguchi H, Omoto H, Hanawa T, Minami T. Go-rei-San, a Kampo medicine, reduces postoperative nausea and vomiting: a prospective, single-blind, randomized trial. J Altern Complement Med. 2013 Dec;19(12):946-50. doi: 10.1089/acm.2013.0118. Epub 2013 Jul 9. PMID 23837690
- [Background] Lin KY, Hu YT, Chang KJ, Lin HF, Tsauo JY. Effects of yoga on psychological health, quality of life, and physical health of patients with cancer: a meta-analysis. Evid Based Complement Alternat Med. 2011;2011:659876. doi: 10.1155/2011/659876. Epub 2011 Mar 9. PMID 21437197
- [Background] Maghami M, Afazel MR, Azizi-Fini I, Maghami M. The effect of aromatherapy with peppermint essential oil on nausea and vomiting after cardiac surgery: A randomized clinical trial. Complement Ther Clin Pract. 2020 Aug;40:101199. doi: 10.1016/j.ctcp.2020.101199. Epub 2020 May 18. PMID 32891278
- [Background] Montazeri AS, Raei M, Ghanbari A, Dadgari A, Montazeri AS, Hamidzadeh A. Effect of herbal therapy to intensity chemotherapy-induced nausea and vomiting in cancer patients. Iran Red Crescent Med J. 2013 Feb;15(2):101-6. doi: 10.5812/ircmj.4392. Epub 2013 Feb 5. PMID 24693415
- [Background] Montgomery GH, Schnur JB, Kravits K. Hypnosis for cancer care: over 200 years young. CA Cancer J Clin. 2013 Jan;63(1):31-44. doi: 10.3322/caac.21165. Epub 2012 Nov 20. PMID 23168491
- [Background] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456
- [Background] Obrink E, Jildenstal P, Oddby E, Jakobsson JG. Post-operative nausea and vomiting: update on predicting the probability and ways to minimize its occurrence, with focus on ambulatory surgery. Int J Surg. 2015 Mar;15:100-6. doi: 10.1016/j.ijsu.2015.01.024. Epub 2015 Jan 29. PMID 25638733
- [Background] Saberi F, Sadat Z, Abedzadeh-Kalahroudi M, Taebi M. Acupressure and ginger to relieve nausea and vomiting in pregnancy: a randomized study. Iran Red Crescent Med J. 2013 Sep;15(9):854-61. doi: 10.5812/ircmj.12984. Epub 2013 Sep 5. PMID 24616799
- [Background] Stallings-Welden LM, Doerner M, Ketchem EL, Benkert L, Alka S, Stallings JD. A Comparison of Aromatherapy to Standard Care for Relief of PONV and PDNV in Ambulatory Surgical Patients. J Perianesth Nurs. 2018 Apr;33(2):116-128. doi: 10.1016/j.jopan.2016.09.001. Epub 2017 Mar 16. PMID 29580591
- [Background] Sahbaz M, Khorshid L. The Effect of Cold Vapor and Ice Cube Absorption in the Early Postoperative Period on Sore Throat and Hoarseness Induced by Intubation. J Perianesth Nurs. 2020 Oct;35(5):518-524. doi: 10.1016/j.jopan.2019.12.007. Epub 2020 May 10. PMID 32402773
- [Background] Weibel S, Rucker G, Eberhart LH, Pace NL, Hartl HM, Jordan OL, Mayer D, Riemer M, Schaefer MS, Raj D, Backhaus I, Helf A, Schlesinger T, Kienbaum P, Kranke P. Drugs for preventing postoperative nausea and vomiting in adults after general anaesthesia: a network meta-analysis. Cochrane Database Syst Rev. 2020 Oct 19;10(10):CD012859. doi: 10.1002/14651858.CD012859.pub2. PMID 33075160
- See also: Aygin, D. (2016). Bulantı ve kusma. Yoğun Bakım Hemşireliği Dergisi, 20(1), 44-56. — https://dergipark.org.tr/en/download/article-file/260207
- See also: Durmaz, M., & Burucu, R. (2019). Ameliyat Sonrası Bulantı ve Kusmayı Önlemede Kullanılan Farmakolojik Olmayan Yöntemlerin Kanıt Düzeyleri. İzmir Katip Çelebi Üniversitesi Sağlık Bilimleri Fakültesi Dergisi, 4(3), 97-104. — https://dergipark.org.tr/en/download/article-file/905335
- See also: Hepkarşı, A., Bor, C., Demirağ, K., Çankayalı, İ., Uyar, M. (2015). Yoğun Bakım Sedasyonunda Ramsay-Richmond Skalaları ve Hemşire-Doktor Arasındaki Uyumun Karşılaştırılması. J Turk Soc Intens Care,13,112-6 doi: 10.4274/tybdd.20592 — https://web.s.ebscohost.com/ehost/pdfviewer/pdfviewer?vid=0&sid=47c3f6b5-3059-480d-9755-8c56d1cb6b8f%40redis
- See also: Irmak, B., & Karadağ, M. Ameliyat sonrası bulantı ve kusmanın yönetiminde aromaterapinin etkisini değerlendiren çalışmaların incelenmesi. Cerrahi Ameliyathane Sterilizasyon Enfeksiyon Kontrol Hemşireliği Dergisi, 2(1), 11-30. — https://dergipark.org.tr/en/download/article-file/1528058
- See also: Jung, M. Y., Choi, H. S., & Park, K. Y. (2012). Effects of Postoperative Oral Care Using Cold Therapy on Nausea, Vomiting and Oral Discomfort in Patients with Laparoscopic Myomectomy. Journal of Korean Academy of Fundamentals of Nursing, 19(3), 292-301. — https://www.koreascience.or.kr/article/JAKO201225841538964.page
- See also: Sözen, K. K. (2020). Ameliyat sonrası derlenme ünitesinde görülen erken dönem komplikasyonlarının değerlendirilmesi. Çukurova Anestezi ve Cerrahi Bilimler Dergisi, 3(3), 212-222. — https://dergipark.org.tr/en/download/article-file/1424225
- See also: Yaman Aktaş, Y., Gürçayır, D., & Atalay, C. (2018). Ameliyat sonrası bulantı kusma yönetiminde kanıta dayalı uygulamalar. Dicle Tıp Dergisi, 45(3), 341-351. — https://dergipark.org.tr/en/download/article-file/530630
- See also: Zaman, F., & Karahan, E. (2020). The Effect of Cold Vapor Treated to Thyroidectomy Patients During Early Postoperative Period. Eastern Journal of Medicine, 25(1), 118-125. — https://jag.journalagent.com/ejm/pdfs/EJM-18189-ORIGINAL_ARTICLE-KARAHAN.pdf